CLINICAL TRIAL: NCT03991104
Title: A Phase I/II Study of S-1 and Oxaliplatin Based Definitive Concurrent Chemoradiotherapy (SOX-CRT-01) for Unresectable Locally Advanced Esophageal Cancer.
Brief Title: SOX-based CRT for Esophageal Cancer.
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No eligible patients enrolled. We have to withdraw the trial.
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yongshi Jia, Head of Radiation Oncology, Zhejiang Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zhejiang Provincal PH006
Record Dates: First submitted 2019-06-15; First posted 2019-06-19 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; chemoradiotherapy; oxaliplatin; S-1
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Oxaliplatin; S 1 (combination); Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SOX-based Chemoradiotherapy (Experimental): IMRT is delivered with a daily fraction of 1.8 Gy to a total dose of 50.4 Gy over 5 weeks. Concurrent Oxaliplatin (3 levels for phase I: 110mg/m², 120 mg/m² and 130 mg/m², d1) and fixed dose of S-1 (80mg/ m², d1-14) are administered concurrently with IMRT, every 4 weeks. The recommended dose of Oxaliplatin are then further evaluated in the Phase II setting.
  Interventions: Drug: Oxaliplatin; Drug: S-1 capsule; Radiation: Intensity modulated radiotherapy (IMRT)

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin (3 levels for phase I: 110 mg/m², 120 mg/m² and 130 mg/m²) is administered as a 2 h intravenous infusion in 500 mL of 5% glucose on day 1 and day 29 during the treatment course.
Drug: S-1 capsule — Patients received a fixed dose of S-1 with a dose of 80 mg/m2/d twice daily for 2 weeks, every 4 weeks.
Radiation: Intensity modulated radiotherapy (IMRT) — The total radiation dose was set to 50.4 Gy, which was given in 28 fractions of 1.8 Gy once-daily fractions for over 5 weeks.

SUMMARY:
Patients with esophageal cancer that had locally advanced diseases or with unresectable diseases are being asked to participate in this phase I/II study.

This phase I/II study is being conducted to determine the maximum-tolerated dose (MTD), dose-limiting toxicity (DLT), and efficacy of IMRT combined with S-1 and Oxaliplatin (SOX) based chemotherapy for unresectable locally advanced esophageal cancer.

DETAILED DESCRIPTION:
Esophageal carcinoma (EC) remains difficult to cure with overall 5-year survival rates for locally advanced stages being poor. Definitive concurrent chemoradiotherapy (dCRT) remains the mainstay of treatment for locally advanced and unresectable EC. Oxaliplatin is a new generation platinum with a more preferable toxicity profile compared to cisplatin. Furthermore, S-1 combines 5-Fu prodrug (tegafur) and two modulators of 5-Fu metabolism, gimeracil (CDHP) and oteracil. Basic studies showed that S-1 has superior anti-cancer effects than 5-Fu and enhances the sensitivity of cancer cells to the effects of radiotherapy. Herein, we designed a prospective phase I/II study, which is combined S-1 and oxaliplatin with IMRT for the patients with locally advanced and unresectable esophageal cancer, and evaluated the tolerability and efficacy of this combination.

<Phase I>

Primary Objective:

To establish the safety of combination chemotherapy comprising oxaliplatin (escalating doses: 110, 120, 130 mg/m2, day 1 and day 29), fixed dose of S-1 (80 mg/m2, day1-14 and day 29-42) and IMRT (5040cGy/28fx/5W+) in unresectable locally advanced esophageal cancer.

Secondary Objective:

To observe the efficacy of this regimen in these patients.

<Phase II>

Primary Objective:

To assess the response rate of combination chemotherapy comprising oxaliplatin (recommended dose determined in phase I study, day1 and day29), fixed dose of S-1 (80 mg/m2, day1-14 and day 29-42), and IMRT (5040cGy/28fx/5W+) in unresectable locally advanced esophageal cancer.

Secondary Objectives:

To determine the adverse reactions of this regimen in these patients. To determine PFS(Progression free survival) of patients treated with this regimen.

To determine OS (overall survival) of patients treated with this regimen. To explore the Health-related Quality of life using EORTC QLQ-C30 and EORTC QLQ-OES18 in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Cytopathological confirmed esophageal cancer with unresectable locally advanced diseases;
2. Age of 18-70;
3. ECOG performance status: 0-1;
4. No treatments prior to enrollment;
5. Patients must have measurable or evaluable disease with at least one tumor mass maximum diameter ≥10mm by multi-slice spiral CT or MR scan. Imaging exam must be performed within 15 days from enrollment.
6. Normal marrow function and the blood tests must be collected within 7 days from enrollment with a hemoglobin of ≥90g/L, an white blood cell (WBC) counts of ≥4.0×109/L，a neutrophil count of ≥2.0×109/L, , a platelet count of ≥100×109/L, a total bilirubin (TBil) of ≤1.0 upper normal limitation (UNL), a creatinine (Cr) of ≤ 1.0 UNL, alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) of ≤2.5 UNL, Alkaline phosphatase (AKP) ≤5.0 UNL. Pulmonary function (FEV1 >1L), and no major electrocardiogram abnormalities.
7. Normal electrocardiogram results and no history of congestive heart failure;
8. Patients must be with good compliance and agree to accept follow-up of disease progression and adverse events;
9. Informed consent signed.

Exclusion Criteria:

1. Prior treatments of chemotherapy or irradiation;
2. Poor bone marrow, liver and kidney functions, which would make chemotherapy intolerable;
3. Contraindication for irradiation: complete obstruction of esophagus, deep esophageal ulcer, fistula to mediastinum, or haematemesis;
4. Participating in other clinical trials;
5. Pregnancy, breast feeding, or not adopting birth control;
6. Clinically significant and uncontrolled major medical conditions including but not limited to: active uncontrolled infection, symptomatic congestive heart failure, Unstable angina pectoris or cardiac arrhythmia, psychiatric illness/ social situation that would limit compliance with study requirements; any medical condition, which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities;
7. Weight loss of 20% or more of normal body weight within 3 months.
8. The subject has had another active malignancy within the past five years except for cervical cancer in site, in situ carcinoma of the bladder or non-melanoma carcinoma of the skin;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 1 month
  Phase I: toxicities will be assessed based on the common toxicity criteria for adverse events version 4.0 (CTCAE v4.0).
Response rate | 1 month
  Phase II: Response rate will be done after 4 weeks following the last radiotherapy session as evaluated by RECIST 1.1.

SECONDARY OUTCOMES:
Recommended dose of Oxaliplatin for phase II trial. | 1 month
  To determine the recommended phase II dose (RD) of Oxaliplatin with fixed dose of S-1 in combination with IMRT for esophageal cancer (Phase I).
Number of Participants with Adverse Events (Phase II). | 6 months
  Both the number of subjects with adverse events and the degree of the adverse events of each participant according to NCI CTCAE version 4.0 will be recorded. And the outcome of each adverse event will be followed.
Overall survival time | 0-2 years
  Overall survival (OS) is determined as the time (in months) between the first day of therapy and the last follow-up or the date of death.
Progression-free survival time | 0-2 years
  Progression-free survival (PFS) is calculated from the date of CRT initiation to the date of documented failure (local recurrence or metastasis occurrence) or the date of the last follow-up for those remaining.

OTHER OUTCOMES:
Health-related Quality of life (HR-QoL, Phase II) | 0-2 years
  In phase II trial, HR-QoL would be measured by standardized EORTC questionaires (EORTC QLQ-C30).
Health-related Quality of life (HR-QoL, Phase II) | 0-2 years
  In phase II trial, HR-QoL would be measured by standardized EORTC questionaires (EORTC QLQ-OES18).

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China